CLINICAL TRIAL: NCT05302453
Title: The Effect of Basic Body Awareness Therapy on Musculoskeletal Disorders and Psychological Symptoms in University Students Participating in the Hybrid Education Program During the COVID-19 Pandemic Process
Brief Title: The Effect of Basic Body Awareness Therapy on Musculoskeletal Disorders and Psychological Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hamiyet Yuce, Assistant Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1
Record Dates: First submitted 2022-03-13; First posted 2022-03-31 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: University Students
Keywords: Basic Body Awareness Therapy; COVID-19; Musculoskeletal Pain; telerehabilitation; mental health
MeSH Terms: conditions — COVID-19; Musculoskeletal Pain; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic Body Awareness Therapy Group (Experimental): BBAT exercises to the participants in the study group, were performed under the leadership of two physiotherapists with internationally valid training certificates. In the face-to-face training, BBAT exercises were taught to the participants. Then the training went on via Google Meet. The lying exercises were shown on one participant before each group study and participants were asked to do lying exercises at home. Sitting and lying exercises were performed as a hybrid at one hour/in a week for 12 weeks. At the beginning and end of each group training, feedback was received from the participants' own experiences of the effects of the exercises on the body, emotions, and thoughts.
  Interventions: Other: Basic Body Awareness Therapy
- Control Group (No Intervention): The Control group was warned to continue with daily routines and not to take any training that includes body-mind approaches such as yoga or Tai chi for 12 weeks.

INTERVENTIONS:
Other: Basic Body Awareness Therapy — Basic Body Awareness Therapy (BBAT), which is among the body-mind approaches, is also frequently used in the rehabilitation of patients with psychiatric disorders, pain, and chronic musculoskeletal system problems.
  Arms: Basic Body Awareness Therapy Group

SUMMARY:
During the coronavirus disease (COVID-19) pandemic, stay-at-home isolation as a precaution to alleviate the disease has affected the physical and mental well-being of individuals. University students spent time in front of the screen with online education and developed a sedentary lifestyle during the academic term. In this process, musculoskeletal disorders increased more in university students due to the increase in the use of laptop or computer, smartphone, and social media. The COVID-19 pandemic has caused psychological disorders as well as physical health problems. General population studies have shown that all forms of depression, anxiety, stress, sleep problems, and psychological distress are highly increased during this period. In a study conducted in Turkey, it was reported that students' negative well-being, anxiety, and physical inactivity significantly affected perceived stress during the COVID-19 pandemic, and students' mental health was at high risk. It has been stated that providing mental health supportive systems in students and encouraging physical activity regularly can reduce perceived stress levels.

On the other hand, psychological interventions via video conferencing platforms have been proposed to promote mental health due to the limited and delayed face-to-face healthcare as a result of the COVID-19 pandemic. It has been stated that the use of telemedicine or e-health applications together with body-mind approaches such as yoga, tai chi, qigong may be beneficial in order to encourage physical activity and protect mental health in this critical period. Basic Body Awareness Therapy (BBAT), which is among the body-mind approaches, is also frequently used in the rehabilitation of patients with psychiatric disorders, pain, and chronic musculoskeletal system problems. Therefore, the aim of this study is to evaluate the effect of BBAT on musculoskeletal disorders and psychological symptoms in university students who participated in the hybrid (online + face-to-face) education program during the COVID-19 pandemic. The importance of this study is that it is the first study on physical and psychological symptoms of BBAT in university students.

ELIGIBILITY:
Inclusion Criteria:

* Being studying at Bandirma Onyedi Eylul University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
* Volunteering to participate in the study
* Being between the ages of 18-25

Exclusion Criteria:

* Having any diagnosed psychological disorder
* Regularly doing body-mind approaches such as yoga and tai chi
* Having any condition involving the musculoskeletal system
* Having a rheumatic disease

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) | Baseline
  The Turkish reliability and validity studies of the questionnaire developed by Cornell University were performed by Erdinc et al. The CMDQ measures the frequency of pain or discomfort in 11 different body parts in the past seven days, the severity of this situation, and its interference on the ability to work.For frequency in scoring the scale: "never: 0 points, 1-2 times last week: 1.5 points, 3-4 times last week: 3.5 points, once every day: 5 points, several times every day: 10 points are taken. For severity: slightly uncomfortable: 1 point, moderately uncomfortable: 2 points, very uncomfortable: 3 points. For the interference on the ability to work: not at all: 1 point, slightly interfered: 2 points, substantially interfered: 3 points. Higher scores mean a worse outcome.
Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) | 12th week
  The Turkish reliability and validity studies of the questionnaire developed by Cornell University were performed by Erdinc et al. The CMDQ measures the frequency of pain or discomfort in 11 different body parts in the past seven days, the severity of this situation, and its interference on the ability to work.For frequency in scoring the scale: "never: 0 points, 1-2 times last week: 1.5 points, 3-4 times last week: 3.5 points, once every day: 5 points, several times every day: 10 points are taken. For severity: slightly uncomfortable: 1 point, moderately uncomfortable: 2 points, very uncomfortable: 3 points. For the interference on the ability to work: not at all: 1 point, slightly interfered: 2 points, substantially interfered: 3 points. Higher scores mean a worse outcome.
Brief Symptom Inventory (BSI) (53 items) | Baseline
  Sahin & Durak found that the inventory developed by Derogatis is valid and reliable in determining the psychological problems of university students. It has been stated that it is a useful inventory in screening studies of university students' mental health. It is a 53-item self-assessment inventory. BSI uses a 5-point Likert scale, ranging from 0 ("not at all") to 4 ("extremely"). Higher scores mean a worse outcome
Brief Symptom Inventory (BSI) (53 items) | 12th week
  Sahin & Durak found that the inventory developed by Derogatis is valid and reliable in determining the psychological problems of university students. It has been stated that it is a useful inventory in screening studies of university students' mental health. It is a 53-item self-assessment inventory. BSI uses a 5-point Likert scale, ranging from 0 ("not at all") to 4 ("extremely"). Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylul University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen B, Sun J, Feng Y. How Have COVID-19 Isolation Policies Affected Young People's Mental Health? - Evidence From Chinese College Students. Front Psychol. 2020 Jun 24;11:1529. doi: 10.3389/fpsyg.2020.01529. eCollection 2020. PMID 32670172
- [Background] Bravo C, Skjaerven LH, Espart A, Guitard Sein-Echaluce L, Catalan-Matamoros D. Basic Body Awareness Therapy in patients suffering from fibromyalgia: A randomized clinical trial. Physiother Theory Pract. 2019 Oct;35(10):919-929. doi: 10.1080/09593985.2018.1467520. Epub 2018 May 3. PMID 29723080
- [Background] Seferiadis A, Ohlin P, Billhult A, Gunnarsson R. Basic body awareness therapy or exercise therapy for the treatment of chronic whiplash associated disorders: a randomized comparative clinical trial. Disabil Rehabil. 2016;38(5):442-51. doi: 10.3109/09638288.2015.1044036. Epub 2015 May 8. PMID 25955823
- [Derived] Yuce H, Kecelioglu S, Akcay B, Yilmaz FN. Effects of basic body awareness therapy via hybrid telerehabilitation on musculoskeletal and psychological symptoms in university students: A single-blind randomized controlled trial. J Back Musculoskelet Rehabil. 2025 Sep 25:10538127251378088. doi: 10.1177/10538127251378088. Online ahead of print. PMID 40997245